CLINICAL TRIAL: NCT01942135
Title: MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PHASE 3 TRIAL OF FULVESTRANT (FASLODEX (REGISTERED)). WITH OR WITHOUT PD-0332991 (PALBOCICLIB) +/- GOSERELIN IN WOMEN WITH HORMONE RECEPTOR-POSITIVE, HER2-NEGATIVE METASTATIC BREAST CANCER WHOSE DISEASE PROGRESSED AFTER PRIOR ENDOCRINE THERAPY
Brief Title: Palbociclib (PD-0332991) Combined With Fulvestrant In Hormone Receptor+ HER2-Negative Metastatic Breast Cancer After Endocrine Failure (PALOMA-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A5481023; 2013-002580-26 (EudraCT Number)
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Palbociclib (PD-0332991); Fulvestrant; Goserelin; Hormone receptor-+; HER2-negative; Prior Endocrine treatment; any menopausal status; PALOMA-3
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Given until objective progression, symptomatic deterioration, unacceptable toxicity, death, or withdrawal of consent, whichever occurs first.
  Interventions: Drug: Palbociclib; Drug: Fulvestrant
- Arm B (Active Comparator): Given until objective progression, symptomatic deterioration, unacceptable toxicity, death, or withdrawal of consent, whichever occurs first.
  Interventions: Drug: Placebo; Drug: Fulvestrant

INTERVENTIONS:
Drug: Palbociclib — Palbociclib 125 mg/day orally continuously dosed for 3 weeks followed by 1 week off; repeated at each subsequent cycle.
  Arms: Arm A
Drug: Fulvestrant — Fulvestrant 500 mg intramuscularly on Days 1 and 15 of Cycle 1, and then on Day 1 of each subsequent 28 day cycle.
  Arms: Arm A
Drug: Placebo — Placebo orally continuously dosed for 3 weeks followed by 1 week off; repeated at each subsequent cycle.
  Arms: Arm B
Drug: Fulvestrant — Fulvestrant 500 mg intramuscularly on Days 1 and 15 of Cycle 1, and then on Day 1 of each subsequent 28 day cycle.
  Arms: Arm B

SUMMARY:
The study is a randomized, double blind, placebo controlled, Phase 3 clinical trial with the primary objective of demonstrating the superiority of palbociclib in combination with fulvestrant (Faslodex®) over fulvestrant alone in prolonging PFS in women with HR+, HER2 negative metastatic breast cancer whose disease has progressed after prior endocrine therapy. The safety between the two treatment arms will also be compared. During study treatment, pre- and perimenopausal women must be receiving therapy with the LHRH agonist goserelin (Zoladex® or generic).

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older with metastatic or locally advanced disease, not amenable to curative therapy
* Confirmed diagnosis of HR+/HER2- breast cancer
* Any menopausal status
* Progressed within 12 months from prior adjuvant or progressed within 1 month from prior advanced/metastatic endocrine breast cancer therapy
* On an LHRH agonist for at least 28 days, if pre-/peri-menopausal, and willing to switch to goserelin (Zoladex ®) at time of randomization.
* Measurable disease defined by RECIST version 1.1, or bone-only disease
* Eastern Cooperative Oncology Group (ECOG) PS 0-1
* Adequate organ and marrow function, resolution of all toxic effects of prior therapy or surgical procedures
* Patient must agree to provide tumor tissue from metastatic tissue at baseline

Exclusion Criteria:

* Prior treatment with any CDK inhibitor, fulvestrant, everolimus, or agent that inhibits the PI3K-mTOR pathway
* Patients with extensive advanced/metastatic, symptomatic visceral disease, or known uncontrolled or symptomatic CNS metastases
* Major surgery or any anti-cancer therapy within 2 weeks of randomization
* Prior stem cell or bone marrow transplantation
* Use of potent CYP3A4 inhibitors or inducers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 521 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2014-12-05 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (239):
- United States (127):
  - University of Alabama at Birmingham, The Kirklin Clinic, Birmingham, Alabama
  - UAB Hospital-Investigational Drug Service, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Southern Cancer Center, PC, Daphne, Alabama
  - Southern Cancer Center, PC, Mobile, Alabama
  - Southern Cancer Center,PC, Mobile, Alabama
  - Arizona Center for Cancer Care, Avondale, Arizona
  - Ironwood Physicians P.C dba Ironwood Cancer & Research Centers, Chandler, Arizona
  - Arizona Oncology Associates, PC- HAL, Flagstaff, Arizona
  - Ironwood Physicians P.C dba Ironwood Cancer & Research Centers, Gilbert, Arizona
  - Palo Verde Hematology Oncology, Glendale, Arizona
  - Arizona Center for Cancer Care, Glendale, Arizona
  - Western Regional Medical Center, Inc., Goodyear, Arizona
  - Ironwood Physicians P.C dba Ironwood Cancer & Research Centers, Mesa, Arizona
  - Arizona Oncology Associates, PC- HAL, Prescott Valley, Arizona
  - Arizona Oncology Associates, PC- HAL, Sedona, Arizona
  - Arizona Center for Cancer Care, Surprise, Arizona
  - The University of Arizona Cancer Center- North Campus, Tucson, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - CBCC Global Research Inc. at Comprehensive Blood and Cancer Center, Bakersfield, California
  - Administrative Management Only: Translational Research Management, Culver City, California
  - City of Hope, Duarte, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - Global Research Management, Glendale, California
  - UC San Diego Medical Center-La Jolla, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Keck Hospital of USC, Los Angeles, California
  - LAC & USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Hematology Oncology, Los Angeles, California
  - Breastlink Medical Group, Inc., Orange, California
  - Hematology Oncology Medical Group of Orange County, Inc. (HOMG), Orange, California
  - The Center for Cancer Prevention and Treatment at St. Joseph Hospital of Orange, Orange, California
  - UCLA Hematology/Oncology - Pasadena, Pasadena, California
  - UC San Diego Medical Center-Hillcrest, San Diego, California
  - University of California, San Francisco: Helen Diller Comprehensive Cancer Center, San Francisco, California
  - San Luis Obispo Oncology and Hematology Health Center/Pacific Central Coast Health Centers, San Luis Obispo, California
  - Breastlink Medical Group, Inc., Santa Ana, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - City of Hope, South Pasadena, California
  - Torrance Health Association, DBA Torrance Memorial Physician Network/Cancer Care Associates, Torrance, California
  - Torrance Memorial Physician Network-Cancer Care, Torrance, California
  - Wellness Oncology & Hematology, West Hills, California
  - UCLA Hematology - Oncology Clinic - Westlake Village, Westlake Village, California
  - ATTN - Research Pharmacist, Aurora, Colorado
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - Mount Sinai Medical Center- Aventura, Aventura, Florida
  - Sylvester Comprehensive Cancer Center Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Hospitals and Clinics (UHMC) Sylvester at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital/Michael and Dianne Bienes Comprehensive Cancer Center, Fort Lauderdale, Florida
  - Memorial Breast Cancer Center at Memorial Regional Hospital, Hollywood, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - University of Miami Hospitals & Clinics, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health, Ocoee, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Memorial Breast Cancer Center at Memorial Hospital West, Pembroke Pines, Florida
  - Memorial Cancer Institute at Memorial Hospital West, Pembroke Pines, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Sylvester at Plantation, Plantation, Florida
  - Piedmont Cancer Institute, PC, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital, Austell, Georgia
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Cartersville, Georgia
  - Piedmont Cancer Institute, PC, Fayetteville, Georgia
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Marietta, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Cancer Treatment Centers of America at Midwestern Regional Medical Center, Zion, Illinois
  - Maine Center for Cancer Medicine, dba: New England Cancer Specialists, Brunswick, Maine
  - Maine Center for Cancer Medicine, dba: New England Cancer Specialists, Kennebunk, Maine
  - Maine Center for Cancer Medicine, dba: New England Cancer Specialists, Scarborough, Maine
  - Sidney Kimmel Comprehensive Cancer Center (SKCCC) at Johns Hopkins, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center (SKCCC) at Johns Hopkins, Green Spring Station, Lutherville, Maryland
  - University of Michigan Health System/Comprehensive Cancer Center, Ann Arbor, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Fairview Southdale Oncology Clinic, Edina, Minnesota
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - University of Minnesota Physicians, Masonic Cancer Center, Minneapolis, Minnesota
  - Mercy Clinic St. Louis Cancer and Breast Institute, Ballwin, Missouri
  - Mercy Ministry Office, Chesterfield, Missouri
  - Mercy Clinic St. Louis Cancer and Breast Institute, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Mercy Hospital St.Louis- David C. Pratt Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - CareMount Medical, Brewster, New York
  - ProHEALTHCARE Associates, LLP, Lake Success, New York
  - CareMount Medical, Mount Kisco, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Hope Women's Cancer Centers, Asheville, North Carolina
  - Mission Hospital, Inc., Asheville, North Carolina
  - UPMC Cancer Center, Monroeville, Monroeville, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, William M. Cooper Pavilion, Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The Jones Clinic, PC, Germantown, Tennessee
  - Texas Oncology- Dallas Presbyterian Hospital, Dallas, Texas
  - Investigational Products Center (IPC), Fort Worth, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - US Oncology lnvestigational Products Center (IPC), Irving, Texas
  - Texas Oncology- Longview Cancer Center, Longview, Texas
  - Texas Oncology- McAllen South Second Street, McAllen, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology- Tyler, Tyler, Texas
  - Texas Oncology- Weslaco, Weslaco, Texas
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, PC, Arlington, Virginia
  - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - Inova Medical Group, Fairfax, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Leesburg, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Shenandoah Oncology, P.C., Winchester, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Medical Center First Hill IDS Pharmacy, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Columbia St. Mary's, Mequon, Wisconsin
  - Columbia St. Mary's, Milwaukee, Wisconsin
- Australia (15):
  - Bankstown - Lidcombe Hospital, Bankstown, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - River City Pharmacy, Auchenflower, Queensland
  - Sunshine Coast Hospital and Health Service, Nambour, Queensland
  - Icon Cancer Care Southport, Southport, Queensland
  - Cabrini Brighton, Brighton, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Peninsula and Southeast Oncology, Frankston, Victoria
  - Barwon Health, University Hospital Geelong, Geelong, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Peter MacCallum Cancer Centre Pharmacy, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sunshine Hospital Clinical Trials Pharmacy, St Albans, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Fiona Stanley Hospital - Cancer Centre, Murdoch, Western Australia
- Belgium (13):
  - UZ Antwerpen, Edegem, Antwerpen
  - Clinique Saint-Pierre, Ottignies, Brabant Wallon
  - Institut Jules Bordet, Brussels, Brussels Capital
  - Grand Hôpital de Charleroi - Site Notre Dame, Charleroi, Hainaut
  - INDC Entité Jolimontoise - CH de Jolimont-Lobbes, Haine-Saint-Paul, Hainaut
  - CHWaPi - Site IMC, Tournai, Hainaut
  - C.H. de l'Ardenne - site Libramont, Libramont-Chevigny, Luxembourg
  - Hopital Erasme, Brussels, Region de Bruxelles-capital
  - Imelda Ziekenhuis, Bonheiden
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven - Campus Gasthuisberg, Leuven
  - CHU UCL Namur - Site Sainte-Elisabeth, Namur
  - GZA Ziekenhuizen - Campus St Augustinus, Wilrijk
- Canada (11):
  - British Columbia Cancer Agency - Sindi Ahluwalia Hawkins Centre for the Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency - Fraser Valley Centre, Surrey, British Columbia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Cancer Centre of Southeastern Ontario @ Kingston Health Sciences Centre, Kingston, Ontario
  - Lakeridge Health Oshawa, R.S. McLaughlin Durham Regional Cancer Centre, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre, General Campus, Ottawa, Ontario
  - Niagara Health System Walker Family Cancer Center, St. Catharines, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Germany (3):
  - Universitaetsklinikum Leipzig AoeR, Leipzig
  - Zentrum fuer Radiologie und Nuklearmedizin am Johannisplatz, Leipzig
  - Klinikum der Universität München, München
- Bon Secours Hospital, Cork, Ireland
- Italy (17):
  - Azienda Sanitaria Firenze, c/o Ospedale S. M. Annunziata Farmacia Interna, Bagno A Ripoli (FI)
  - S.O.C. Oncologia Medica I, Azienda Sanitaria Firenze, c/o Ospedale S. M. Annunziata, Bagno A Ripoli (FI)
  - SSD Oncologia Medica Addarii-Zamagni A.O.U. di Bologna Policlinico S. Orsola Malpighi, Bologna
  - U.O. di Oncologia Medica P.O. Policlinico G. Rodolico", Catania
  - Azienda U.L.S.S. n. 21 di Legnago, Presidio Ospedaliero Mater Salutis, Legnago (VR)
  - Farmacia Ospedaliera-Azienda U.L.S.S. n. 21 di Legnago, Legnago (VR)
  - IRST, Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola (FC)
  - Farmacia IRCCS Ospedale San Raffaele, Milan
  - IRCCS Ospedale S. Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Servizio di Farmacia - Istituto Europeo di Oncologia, Milan
  - Policlinico di Modena Dipartimento ad attivita integrata di Oncologia,, Modena
  - IRCCS Istituto Nazionale per lo Studio e la Cura dei Tumori, Napoli
  - Farmacia - Fondazione Policlinico Universitario A. Gemelli, Roma
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - S.C. Oncologia, A.O.S. Maria, Terni
- Japan (8):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Saitama Cancer Center, Kita-adachi-gun, Saitama,japan
  - Chiba Cancer Center, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hakuaikai Medical Corporation Sagara Hospital, Kagoshima
  - National Hospital Organization, Osaka
- Netherlands (6):
  - Academisch Ziekenhuis Maastricht, Maastricht, Limburg
  - Orbis Medisch Centrum, Sittard-Geleen, Limburg
  - TweeSteden Ziekenhuis, Tilburg, North Brabant
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Ikazia Ziekenhuis, Rotterdam, South Holland
  - Haga Ziekenhuis, The Hague, South Holland
- Portugal (2):
  - Champalimaud Cancer Center/ Breast Unit, Lisbon
  - Instituto Português de Oncologia, Porto
- Romania (4):
  - Spitalul Clinic CF nr.2 Bucuresti, Bucharest
  - Spitalul Municipal Ploiesti, Ploieşti
  - Spitalul Judetean de Urgente "Sf. Ioan cel Nou", Suceava
  - Spitalul Clinic Judetean Mures, Tg. Mures
- Russia (12):
  - GBUZ Republican Clinical Oncology Dispensary of Ministry of Health of the Republic of Bashkortostan, Ufa, Bashkortostan Republic
  - OGBUZ Belgorod Oncology Dispensary, Belgorod, Belgorod Oblast
  - OGBUZ Belgorod Oncology Dispensary, Stariy Oskol, Belgorod Oblast
  - GBUZ Leningrad regional oncological dispensary, Village Kuzmolovsky, Leningradskaya Oblast'
  - FGBUZ Clinical Hospital 101 of the Federal Medical and Biological Agency", Lermontov, Stavropol Territory
  - GBUZ of Stavropol Territory "Pyatigorsk Oncology Dispensary", Pyatigorsk, Stavropol Territory
  - GBUZ Chelyabinsk regional clinical center of oncology and nuclear medicine, Chelyabinsk
  - FSBSI Russian Cancer Research Center n.a.NN Blokhin, Moscow
  - Saint Petersburg GBUZ "City Clinical Oncology Dispensary", Saint Petersburg
  - Saint Petersburg GBUZ City Clinical Oncology Dispensary, Saint Petersburg
  - GBUZ of Stavropol Territory "Stavropol Regional Clinical Oncology Dispensary", Stavropol
  - FGBU Russian Research Center for Radiology and Surgical Technologies, Village Pesochny
- South Korea (5):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Asan medical Center, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Ege University Medical Faculty, Izmir, Bornova, Turkey (Türkiye)
- Ukraine (6):
  - Oblasne komunalne nekomertsiine pidpryiemstvo "Bukovynskyi klinichnyi onkolohichnyi tsentr", Chernivtsi
  - Komunalnyi zaklad 'Miska klinichna likarnia No.4' Dniprovskoi miskoi rady,, Dnipro
  - Komunalne nekomertsiyne pidpryiemstvo "Oblasnyi, Kharkiv
  - KNP Lvivskoi oblasnoi rady Lvivskyi onkolohichnyi, Lviv
  - Komunalna ustanova "Odeska oblasna klinichna likarnia", Odesa
  - Podilskyi rehionalnyi tsentr onkolohii,, Vinnytsia
- United Kingdom (6):
  - Queen Alexandra Hospital, Portsmouth Hospitals NHS Trust Portsmouth Haematology and Oncology Centre, Portsmouth, Hampshire
  - Velindre Cancer Centre, Cardiff, South Glamorgan
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - Sheffield Teaching Hospitals NHS Foundation Trust, Weston Park Hospital, Sheffield, South Yorkshire
  - The Royal Marsden NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Li H, Wu Y, Zou H, Koner S, Plichta JK, Tolaney SM, Zhang J, He YW, Wei Q, Tang L, Zhang H, Zhang B, Guo Y, Chen X, Li K, Lian L, Ma F, Luo S. Clinical efficacy of CDK4/6 inhibitor plus endocrine therapy in HR-positive/HER2-0 and HER2-low-positive metastatic breast cancer: a secondary analysis of PALOMA-2 and PALOMA-3 trials. EBioMedicine. 2024 Jul;105:105186. doi: 10.1016/j.ebiom.2024.105186. Epub 2024 Jun 10. PMID 38861871
- [Derived] Rugo HS, Im SA, Joy AA, Shparyk Y, Walshe JM, Sleckman B, Loi S, Theall KP, Kim S, Huang X, Bananis E, Mahtani R, Finn RS, Dieras V. Effect of palbociclib plus endocrine therapy on time to chemotherapy across subgroups of patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative advanced breast cancer: Post hoc analyses from PALOMA-2 and PALOMA-3. Breast. 2022 Dec;66:324-331. doi: 10.1016/j.breast.2022.11.005. Epub 2022 Nov 15. PMID 36463643
- [Derived] Zhu Z, Turner NC, Loi S, Andre F, Martin M, Dieras V, Gelmon KA, Harbeck N, Zhang C, Cao JQ, Yan Z, Lu DR, Wei P, VanArsdale TL, Rejto PA, Huang X, Rugo HS, Loibl S, Cristofanilli M, Finn RS, Liu Y. Comparative biomarker analysis of PALOMA-2/3 trials for palbociclib. NPJ Precis Oncol. 2022 Aug 16;6(1):56. doi: 10.1038/s41698-022-00297-1. PMID 35974168
- [Derived] Rugo HS, Cristofanilli M, Loibl S, Harbeck N, DeMichele A, Iwata H, Park YH, Brufsky A, Theall KP, Huang X, McRoy L, Bananis E, Turner NC. Prognostic Factors for Overall Survival in Patients with Hormone Receptor-Positive Advanced Breast Cancer: Analyses From PALOMA-3. Oncologist. 2021 Aug;26(8):e1339-e1346. doi: 10.1002/onco.13833. Epub 2021 Jun 12. PMID 34037282
- [Derived] Iwata H, Umeyama Y, Liu Y, Zhang Z, Schnell P, Mori Y, Fletcher O, Marshall JC, Johnson JG, Wood LS, Toi M, Finn RS, Turner NC, Bartlett CH, Cristofanilli M. Evaluation of the Association of Polymorphisms With Palbociclib-Induced Neutropenia: Pharmacogenetic Analysis of PALOMA-2/-3. Oncologist. 2021 Jul;26(7):e1143-e1155. doi: 10.1002/onco.13811. Epub 2021 Jun 7. PMID 33955129
- [Derived] Finn RS, Rugo HS, Gelmon KA, Cristofanilli M, Colleoni M, Loi S, Schnell P, Lu DR, Theall KP, Mori A, Gauthier E, Bananis E, Turner NC, Dieras V. Long-Term Pooled Safety Analysis of Palbociclib in Combination with Endocrine Therapy for Hormone Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: Updated Analysis with up to 5 Years of Follow-Up. Oncologist. 2021 May;26(5):e749-e755. doi: 10.1002/onco.13684. Epub 2021 Mar 10. PMID 33486783
- [Derived] Finn RS, Cristofanilli M, Ettl J, Gelmon KA, Colleoni M, Giorgetti C, Gauthier E, Liu Y, Lu DR, Zhang Z, Bartlett CH, Slamon DJ, Turner NC, Rugo HS. Treatment effect of palbociclib plus endocrine therapy by prognostic and intrinsic subtype and biomarker analysis in patients with bone-only disease: a joint analysis of PALOMA-2 and PALOMA-3 clinical trials. Breast Cancer Res Treat. 2020 Nov;184(1):23-35. doi: 10.1007/s10549-020-05782-4. Epub 2020 Aug 11. PMID 32783178
- [Derived] Ettl J, Im SA, Ro J, Masuda N, Colleoni M, Schnell P, Bananis E, Lu DR, Cristofanilli M, Rugo HS, Finn RS. Hematologic adverse events following palbociclib dose reduction in patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative advanced breast cancer: pooled analysis from randomized phase 2 and 3 studies. Breast Cancer Res. 2020 Mar 12;22(1):27. doi: 10.1186/s13058-020-01263-0. PMID 32164785
- [Derived] Masuda N, Mukai H, Inoue K, Rai Y, Ohno S, Mori Y, Hashigaki S, Muramatsu Y, Umeyama Y, Iwata H, Toi M. Neutropenia management with palbociclib in Japanese patients with advanced breast cancer. Breast Cancer. 2019 Sep;26(5):637-650. doi: 10.1007/s12282-019-00970-7. Epub 2019 May 24. PMID 31127500
- [Derived] Turner NC, Liu Y, Zhu Z, Loi S, Colleoni M, Loibl S, DeMichele A, Harbeck N, Andre F, Bayar MA, Michiels S, Zhang Z, Giorgetti C, Arnedos M, Huang Bartlett C, Cristofanilli M. Cyclin E1 Expression and Palbociclib Efficacy in Previously Treated Hormone Receptor-Positive Metastatic Breast Cancer. J Clin Oncol. 2019 May 10;37(14):1169-1178. doi: 10.1200/JCO.18.00925. Epub 2019 Feb 26. PMID 30807234
- [Derived] Masuda N, Inoue K, Nakamura R, Rai Y, Mukai H, Ohno S, Hara F, Mori Y, Hashigaki S, Muramatsu Y, Nagasawa T, Umeyama Y, Huang X, Iwata H. Palbociclib in combination with fulvestrant in patients with hormone receptor-positive, human epidermal growth factor receptor 2-negative advanced breast cancer: PALOMA-3 subgroup analysis of Japanese patients. Int J Clin Oncol. 2019 Mar;24(3):262-273. doi: 10.1007/s10147-018-1359-3. Epub 2018 Nov 3. PMID 30392115
- [Derived] Turner NC, Slamon DJ, Ro J, Bondarenko I, Im SA, Masuda N, Colleoni M, DeMichele A, Loi S, Verma S, Iwata H, Harbeck N, Loibl S, Andre F, Puyana Theall K, Huang X, Giorgetti C, Huang Bartlett C, Cristofanilli M. Overall Survival with Palbociclib and Fulvestrant in Advanced Breast Cancer. N Engl J Med. 2018 Nov 15;379(20):1926-1936. doi: 10.1056/NEJMoa1810527. Epub 2018 Oct 20. PMID 30345905
- [Derived] Cristofanilli M, DeMichele A, Giorgetti C, Turner NC, Slamon DJ, Im SA, Masuda N, Verma S, Loi S, Colleoni M, Theall KP, Huang X, Liu Y, Bartlett CH. Predictors of prolonged benefit from palbociclib plus fulvestrant in women with endocrine-resistant hormone receptor-positive/human epidermal growth factor receptor 2-negative metastatic breast cancer in PALOMA-3. Eur J Cancer. 2018 Nov;104:21-31. doi: 10.1016/j.ejca.2018.08.011. Epub 2018 Oct 8. PMID 30308388
- [Derived] Rugo HS, Turner NC, Finn RS, Joy AA, Verma S, Harbeck N, Masuda N, Im SA, Huang X, Kim S, Sun W, Iyer S, Schnell P, Bartlett CH, Johnston S. Palbociclib plus endocrine therapy in older women with HR+/HER2- advanced breast cancer: a pooled analysis of randomised PALOMA clinical studies. Eur J Cancer. 2018 Sep;101:123-133. doi: 10.1016/j.ejca.2018.05.017. Epub 2018 Jul 25. PMID 30053671
- [Derived] Dieras V, Rugo HS, Schnell P, Gelmon K, Cristofanilli M, Loi S, Colleoni M, Lu DR, Mori A, Gauthier E, Huang Bartlett C, Slamon DJ, Turner NC, Finn RS. Long-term Pooled Safety Analysis of Palbociclib in Combination With Endocrine Therapy for HR+/HER2- Advanced Breast Cancer. J Natl Cancer Inst. 2019 Apr 1;111(4):419-430. doi: 10.1093/jnci/djy109. PMID 30032196
- [Derived] Wedam SB, Beaver JA, Amiri-Kordestani L, Bloomquist E, Tang S, Goldberg KB, Sridhara R, Ibrahim A, Kim G, Kluetz P, McKee A, Pazdur R. US Food and Drug Administration Pooled Analysis to Assess the Impact of Bone-Only Metastatic Breast Cancer on Clinical Trial Outcomes and Radiographic Assessments. J Clin Oncol. 2018 Apr 20;36(12):1225-1231. doi: 10.1200/JCO.2017.74.6917. Epub 2018 Mar 9. PMID 29522361
- [Derived] Turner NC, Finn RS, Martin M, Im SA, DeMichele A, Ettl J, Dieras V, Moulder S, Lipatov O, Colleoni M, Cristofanilli M, Lu DR, Mori A, Giorgetti C, Iyer S, Bartlett CH, Gelmon KA. Clinical considerations of the role of palbociclib in the management of advanced breast cancer patients with and without visceral metastases. Ann Oncol. 2018 Mar 1;29(3):669-680. doi: 10.1093/annonc/mdx797. PMID 29342248
- [Derived] Loibl S, Turner NC, Ro J, Cristofanilli M, Iwata H, Im SA, Masuda N, Loi S, Andre F, Harbeck N, Verma S, Folkerd E, Puyana Theall K, Hoffman J, Zhang K, Bartlett CH, Dowsett M. Palbociclib Combined with Fulvestrant in Premenopausal Women with Advanced Breast Cancer and Prior Progression on Endocrine Therapy: PALOMA-3 Results. Oncologist. 2017 Sep;22(9):1028-1038. doi: 10.1634/theoncologist.2017-0072. Epub 2017 Jun 26. PMID 28652278
- [Derived] Verma S, Bartlett CH, Schnell P, DeMichele AM, Loi S, Ro J, Colleoni M, Iwata H, Harbeck N, Cristofanilli M, Zhang K, Thiele A, Turner NC, Rugo HS. Palbociclib in Combination With Fulvestrant in Women With Hormone Receptor-Positive/HER2-Negative Advanced Metastatic Breast Cancer: Detailed Safety Analysis From a Multicenter, Randomized, Placebo-Controlled, Phase III Study (PALOMA-3). Oncologist. 2016 Oct;21(10):1165-1175. doi: 10.1634/theoncologist.2016-0097. Epub 2016 Jul 1. PMID 27368881
- [Derived] Fribbens C, O'Leary B, Kilburn L, Hrebien S, Garcia-Murillas I, Beaney M, Cristofanilli M, Andre F, Loi S, Loibl S, Jiang J, Bartlett CH, Koehler M, Dowsett M, Bliss JM, Johnston SR, Turner NC. Plasma ESR1 Mutations and the Treatment of Estrogen Receptor-Positive Advanced Breast Cancer. J Clin Oncol. 2016 Sep 1;34(25):2961-8. doi: 10.1200/JCO.2016.67.3061. Epub 2016 Jun 6. PMID 27269946
- [Derived] Harbeck N, Iyer S, Turner N, Cristofanilli M, Ro J, Andre F, Loi S, Verma S, Iwata H, Bhattacharyya H, Puyana Theall K, Bartlett CH, Loibl S. Quality of life with palbociclib plus fulvestrant in previously treated hormone receptor-positive, HER2-negative metastatic breast cancer: patient-reported outcomes from the PALOMA-3 trial. Ann Oncol. 2016 Jun;27(6):1047-1054. doi: 10.1093/annonc/mdw139. Epub 2016 Mar 30. PMID 27029704
- [Derived] Cristofanilli M, Turner NC, Bondarenko I, Ro J, Im SA, Masuda N, Colleoni M, DeMichele A, Loi S, Verma S, Iwata H, Harbeck N, Zhang K, Theall KP, Jiang Y, Bartlett CH, Koehler M, Slamon D. Fulvestrant plus palbociclib versus fulvestrant plus placebo for treatment of hormone-receptor-positive, HER2-negative metastatic breast cancer that progressed on previous endocrine therapy (PALOMA-3): final analysis of the multicentre, double-blind, phase 3 randomised controlled trial. Lancet Oncol. 2016 Apr;17(4):425-439. doi: 10.1016/S1470-2045(15)00613-0. Epub 2016 Mar 3. PMID 26947331
- [Derived] Turner NC, Ro J, Andre F, Loi S, Verma S, Iwata H, Harbeck N, Loibl S, Huang Bartlett C, Zhang K, Giorgetti C, Randolph S, Koehler M, Cristofanilli M; PALOMA3 Study Group. Palbociclib in Hormone-Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2015 Jul 16;373(3):209-19. doi: 10.1056/NEJMoa1505270. Epub 2015 Jun 1. PMID 26030518
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481023&StudyName=Palbociclib%20%28PD-0332991%29%20Combined%20With%20Fulvestrant%20In%20Hormone%20Receptor+%20HER2-Negative%20Metastatic%20Breast%20Cancer%20After%20Endocrine%20Failure%20%28PA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 144 sites in 17 countries that randomized 521 participants. Eligible participants were to have histologically or cytologically proven diagnosis of adenocarcinoma of the breast with evidence of recurrent (local or metastatic) disease.
Pre-assignment Details: The study consisted of a screening visit within 28 days before randomization, an active treatment phase, divided in cycles of 28 days each, and a post-treatment follow-up period during which survival and new anti-cancer therapy information was collected every 3 months for the first 9 months, then every 6 months from the last dose of study intervention.
Groups:
- Palbociclib + Fulvestrant: Participants were administered an initial dose of 125 mg per day orally continuously for 3 weeks followed by 1 week off that can be reduced to 100 mg or 75 mg in case of toxicity; repeated at each subsequent cycle and fulvestrant 500 mg intramuscularly on days 1 and 15 of cycle 1 and then every 28 days. Pre- and perimenopausal women received goserelin at least 4 weeks before study treatment start and continued receiving concurrent ovarian function suppression with goserelin administered subcutaneously every 28 days during the active treatment phase. Maximum treatment duration was 105 cycles.
- Placebo + Fulvestrant: Participants were administered placebo orally continuously dosed for 3 weeks followed by 1 week off; repeated at each subsequent cycle and Fulvestrant 500 mg intramuscularly on Days 1 and 15 of cycle 1 and then every 28 days. Pre- and perimenopausal women received goserelin at least 4 weeks before study treatment start and continued receiving concurrent ovarian function suppression with goserelin administered subcutaneously every 28 days during the active treatment phase. Maximum treatment duration was 93 cycles.
Period: Overall Study
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Started | 347 | 174
Treated | 345 | 172
Completed | 0 | 0
Not Completed | 347 | 174
Not completed — Adverse Event | 21 | 7
Not completed — Global Deterioration of Health Status | 9 | 6
Not completed — Randomized Not Treated | 2 | 2
Not completed — Death | 2 | 1
Not completed — Objective Progression or Relapse + Progressive Disease | 279 | 148
Not completed — Participant Refused to Continue Treatment for Reason Other than Adverse Event | 10 | 3
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 19 | 4

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population or full analysis set included all participants who were randomized, with study intervention assignment designated according to initial randomization, regardless of whether participants received study intervention or received a different drug from that to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant | Total
Number analyzed (Participants) | 347 | 174 | 521
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (11.7) | 56.8 (10.4) | 56.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 347 | 174 | 521
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 11 | 28
  Not Hispanic or Latino | 329 | 161 | 490
  Unknown or Not Reported | 1 | 2 | 3
Menopausal Status [Count of Participants; unit: Participants]
  Postmenopausal | 275 | 138 | 413
  Pre/Perimenopausal | 72 | 36 | 108

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Assessed by the Investigator
Description: PFS is the time from the date of randomization to the date of the first documentation of objective progression of disease (PD)or death due to any cause in absence of documented PD. Participants lacking an evaluation of tumor response after randomization had their PFS time censored on the date of randomization with the duration of a day. Participants with documentation of PD or death after a long interval (2 or more incomplete or non-evaluable assessments) since the last tumor assessment were censored at the time of last objective assessment that did not show PD. The length of PFS was calculated as PFS time (months) =[progression/death date(censor date) - randomization date + 1]/30.4. Progression is defined using Response Evaluation Criteria in Solid Tumors(RECIST v1.1) a 20% increase in the sum of diameters of target lesions and the sum must also demonstrate an absolute increase of at least 5mm or unequivocal progression of existing non-target lesions or the appearance of new lesions.
Time Frame: From randomization date to date of first documentation of progression or death (assessed up to 12 months)
Population: The intent-to-treat (ITT) population or full analysis set included all participants who were randomized, with study intervention, regardless of whether participants received the study intervention or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 347 | 174
months | 9.2 [7.5 to NA] — Not estimable based on the Brookmeyer and Crowley method, because of insufficient number of participants with events. | 3.8 [3.5 to 5.5]
Statistical Analysis 1: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; The primary hypothesis to be tested was H0: λ≥1 versus. HA: λ<1, where λ was the palbociclib plus fulvestrant: placebo plus fulvestrant hazard ratio (HR). A HR less than 1 indicates a reduction in hazard rate in favor of Palbociclib + Fulvestrant. The study was planned to have 90% power and control the type-I error rate at 0.025; Test type: Superiority or Other; p < 0.000001, Stratified Log Rank Test (1-sided) — The overall Type-I error rate was persevered at 1-sided 0.025 level for the analysis of the primary endpoint PFS by the Haybittle-Peto efficacy boundary. The priori threshold for statistical significance was 0.00135; The log rank test stratified by sensitivity to prior hormonal therapy and the presence of visceral metastases based on the randomization information; Hazard Ratio (HR) = 0.422, 95% CI 2-sided [0.318 to 0.560] — Assuming proportional hazards, a hazard ratio less than 1 indicates a reduction in hazard rate in favor of the palbociclib plus fulvestrant arm

2. Secondary Outcome: Overall Survival (OS)-Number of Participants Who Died
Description: OS is defined as the time from date of randomization to date of death due to any cause. In the absence of confirmation of death, survival time was censored to last date the participant was known to be alive. For participants lacking survival data beyond the date of their last follow-up, the OS time was censored on the last date they were known to be alive. Participants lacking survival data beyond randomization were to have their OS times be censored at randomization. The length of OS was calculated as OS time (months) = [death date (censor date) - randomization date + 1]/30.4.
Time Frame: From randomization until death (up to 4.5 years)
Population: The ITT population or full analysis set included all participants who were randomized, with study intervention, regardless of whether participants received the study intervention or received a different drug from that to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 347 | 174
Participants | 201 | 109

3. Secondary Outcome: Overall Survival (OS)
Description: as for outcome 2
Time Frame: From randomization until death (up to 4.5 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 347 | 174
months | 34.9 [28.8 to 40.0] | 28.0 [23.6 to 34.6]
Statistical Analysis 1: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0429, Stratified Log Rank Test (1-sided) — 1-sided p-value from the log-rank test stratified by the presence of visceral metastases and sensitivity to prior endocrine therapy per randomization; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.814, 95% CI 2-sided [0.644 to 1.029] — Assuming proportional hazards, a hazard ratio less than 1 indicates a reduction in hazard rate in favor of palbociclib plus fulvestrant

4. Secondary Outcome: Survival Probabilities at Year 1, Year 2, and Year 3
Description: One-, Two- or Three-year Survival Probability is defined as the probability of survival 1 year, 2 or 3 years after the date of randomization based on the Kaplan-Meier estimate. Survival time was censored to last date the participant is known to be alive.
Time Frame: From randomization until death (assessed up to 36 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Survival Probability
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 347 | 174
Survival Probability
  Survival Probability at Year 1 | 85.5 [81.3 to 88.9] | 84.8 [78.3 to 89.4]
  Survival Probability at Year 2 | 65.3 [59.9 to 70.2] | 57.3 [49.2 to 64.6]
  Survival Probability at Year 3 | 49.6 [44.0 to 54.9] | 40.8 [32.9 to 48.5]

5. Secondary Outcome: Objective Response (OR)
Description: OR is defined as the overall complete response (CR) or partial response (PR) according to the RECIST version 1.1 Objective Response Rate (ORR) is defined as the proportion of participants with CR or PR relative to all randomized participants and randomized participants with measurable disease at baseline. Participants who do not have on-study radiographic tumor re-evaluation, who received anti-tumor treatment other than the study medication prior to reaching a CR or PR, or who died, progressed, or dropped out for any reason prior to reaching a CR or PR were counted as non-responders in the assessment of ORR. Per response evaluation criteria in solid tumors criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), ≥30% decrease in the sum of the longest diameter of target lesions (longest for non-nodal and short axis for nodal target lesions); Overall Response (OR) = CR + PR.
Time Frame: From randomization until end of treatment (assessed up to 2 years)
Population: The ITT population or full analysis set included all participants who were randomized, with study intervention, regardless of whether participants received the study intervention or received a different drug from that to which they were randomized. Randomized participants with measurable disease at baseline was also included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 347 | 174
percentage of participants | 21.0 [16.9 to 25.7] | 8.6 [4.9 to 13.8]
Statistical Analysis 1: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; The exact test is testing the null hypothesis that the odds ratio of objective response rate is less than or equal to 1 vs. the alternative hypothesis that the odds ratio of objective response rate is greater than 1. An Odds Ratio >1 means better response in favor of palbociclib plus fulvestrant arm; Test type: Superiority or Other; p = 0.0001, Exact test (1-sided) — The p-value was not adjusted for multiple comparisons. The priori threshold for statistical significance is 1-sided, alpha=0.025; The 1-sided p-value is from the stratified exact test; Odds Ratio (OR) = 2.783, 95% CI 2-sided [1.563 to 5.603] — An Odds Ratio >1 means better response in favor of the palbociclib plus fulvestrant arm

6. Secondary Outcome: Duration of Response (DR)
Description: DR is defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of disease progression or to death due to any cause, whichever occurs first. If tumor progression data included more than 1 date, the first date was used. DR was calculated as [the date response ended (ie, date of PD or death) - first CR or PR date + 1)]/30.4. Kaplan-Meier estimate of median of the DR is provided below. No inferential statistical analysis were done for DR. The DR was only calculated for the participants with a CR or PR.
Time Frame: From randomization until end of treatment (assessed up to 2 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 347 | 174
Months | 10.4 [8.3 to NA] — Due to less follow up time and insufficient number of participants having duration response. | 9.0 [5.6 to NA] — Due to less follow up time and insufficient number of participants having duration response.

7. Secondary Outcome: Clinical Benefit Response (CBR)
Description: CBR is defined as the overall complete response (CR), partial response (PR) , or stable disease (SD) ≥24 weeks according to the RECIST version 1.1. Clinical Benefit Response Rate (CBRR) is defined as the proportion of participants with CR, PR, or SD ≥24 weeks relative to all randomized participants and randomized participants with measurable disease at baseline. Participants who do not have on-study radiographic tumor re-evaluation, who received antitumor treatment other than the study medication prior to reaching a CR or PR, a best response of SD ≥24 weeks, or who died, progressed, or dropped out for any reason prior to reaching a CR or PR and a best response of SD ≥24 weeks was counted as non-responders in the assessment of CBR. Per RECIST v1.1 for target lesions and assessed by MRI: CR, disappearance of all target lesions; PR, ≥30% decrease in the sum of the longest diameter of target lesions; OR = CR + PR.
Time Frame: From randomization until end of treatment (assessed up to 2 years)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 347 | 174
percentage of participants | 66.3 [61.0 to 71.2] | 39.7 [32.3 to 47.3]
Statistical Analysis 1: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Exact test (1-sided) — [p-value comment as in outcome 5, analysis 1]; The 1-sided p-value is from the stratified exact test; Odds Ratio (OR) = 3.016, 95% CI 2-sided [2.046 to 4.565] — An odds ratio > 1 means better clinical benefit response in favor of palbociclib plus fulvestrant arm

8. Secondary Outcome: Observed Plasma Trough Concentration (Ctrough) for Palbociclib
Description: Ctrough was defined as steady-state predose concentration. Observed directly from data. For palbociclib, a steady-state trough was to be defined as a predose plasma concentration following at least 8 consecutive days of 125 mg daily dose without dosing interruption and the time window for the PK collection was to be between 22 and 26 hours after the dose (the day prior to PK collection) and no more than 1 hour post-dose on the day of PK collection.
Time Frame: Cycle 1/Day 15 and Cycle 2/Day 15
Population: The participants who were treated with Palbociclib + fulvestrant (with or without goserelin) or placebo + fulvestrant (with or without goserelin) and have at least one measured plasma drug concentration. The geometric mean and coefficient of variation was not estimable for Cycle 1/Day 15 and Cycle 2/Day 15 for the reporting arm placebo plus fulvestrant.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 325
nanograms per milliliter (ng/mL)
  Cycle 1/Day 15: number analyzed (Participants) | 165
  Cycle 1/Day 15 | 70.70 (44)
  Cycle 2/Day 15: number analyzed (Participants) | 160
  Cycle 2/Day 15 | 75.29 (44)

9. Secondary Outcome: Ctrough for Fulvestrant
Description: Ctrough was defined as steady-state predose concentration. Observed directly from data. For fulvestrant, a steady-state trough was to be defined when a patient had received all prior planned doses and the sample was collected predose.
Time Frame: Cycles 2/Day 1 and Cycle 3/Day 1
Population: The 40 participants who participated in the early safety review, who are treated with palbociclib + fulvestrant ± goserelin or placebo + fulvestrant ± goserelin and have at least one measured plasma drug concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 64 | 33
ng/mL
  Cycle 2/Day 1: number analyzed (Participants) | 35 | 19
  Cycle 2/Day 1 | 11.75 (41) | 9.31 (52)
  Cycle 3/Day 1: number analyzed (Participants) | 29 | 14
  Cycle 3/Day 1 | 9.90 (42) | 7.60 (72)

10. Secondary Outcome: Ctrough for Goserelin
Description: Ctrough was defined as steady-state predose concentration. Observed directly from data. For goserelin, a steady-state trough was to be defined when a patient had received all prior planned doses and the sample was collected predose.
Time Frame: Cycles 2/ Day 1 and Cycle 3/ Day 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter (pg/mL)
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 16 | 8
picograms per milliliter (pg/mL)
  Cycle 2/Day 1: number analyzed (Participants) | 9 | 5
  Cycle 2/Day 1 | 295.1 (153) | 302.5 (74)
  Cycle 3/Day 1: number analyzed (Participants) | 7 | 3
  Cycle 3/Day 1 | 344.8 (64) | 288.5 (40)

11. Secondary Outcome: Change From Baseline Between Treatment Comparison in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Functional Scale Scores
Description: The EORTC-QLQ-C30 is a 30-item questionnaire composed of five multi-item functional subscales (physical, role, emotional, cognitive , and social functioning), three multi-item symptom scales (fatigue, nausea/vomiting, and pain), a global quality of life (QOL) subscale, and six single item symptom scales assessing other cancer-related symptoms (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and the financial impact of cancer). The questionnaire employs 28 4-point Likert scales with responses from "not at all" to "very much" and two 7-point Likert scales for global health and overall QOL. Responses to all items are then converted to a 0 to 100 scale. For functional and global QOL scales, higher scores represent a better level of functioning/QOL. For symptom-oriented scales, a higher score represents more severe symptoms. A 10-point or higher change in scores from baseline is considered clinically significant.
Time Frame: From Cycle 1 to 14, as of 05 December 2014.
Population: The PRO -evaluable population is defined as a subset of ITT participants, who have completed a baseline and at least one post -baseline PRO assessment prior to end of study treatment. Analysis based on repeated measures mixed-effects model with an intercept term, treatment, time, treatment-by-time, and baseline as covariate.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 335 | 166
Units on a scale
  Global health status / QoL | -0.9 (64.5) [-2.5 to 0.7] | -4.0 (26.25) [-6.3 to -1.7]
  Physical functioning | -0.7 (22.76) [-2.1 to 0.7] | -1.7 (21.24) [-3.7 to 0.2]
  Role functioning | -1.8 (30.70) [-3.7 to 0.1] | -3.7 (28.04) [-6.5 to -0.9]
  Emotional functioning | 2.7 (25.97) [1.1 to 4.3] | -1.9 (21.19) [-4.2 to 0.5]
  Cognitive functioning | -1.7 (20.97) [-3.1 to -0.2] | -2.9 (20.22) [-5.0 to -0.7]
  Social functioning | -0.5 (32.07) [-2.5 to 1.5] | -0.6 (32.27) [-3.4 to 2.3]
Statistical Analysis 1: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for Global health status/ QoL; Test type: Superiority or Other; p = 0.0313, Mixed Model Analysis (2-sided) — The priori threshold for statistical significance is 2-sided alpha=0.05. The p-value was not adjusted for multiple comparisons; Analysis based on repeated measures mixed-effects model with an intercept term, treatment, time, treatment-by-time, and baseline as covariate; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [0.3 to 6.0]
Statistical Analysis 2: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for physical functioning; Test type: Superiority or Other; p = 0.4000, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-1.4 to 3.5]
Statistical Analysis 3: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for role functioning; Test type: Superiority or Other; p = 0.2615, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-1.5 to 5.3]
Statistical Analysis 4: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for emotional functioning; Test type: Superiority or Other; p = 0.0016, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 4.6, 95% CI 2-sided [1.7 to 7.4]
Statistical Analysis 5: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for cognitive functioning; Test type: Superiority or Other; p = 0.3650, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-1.4 to 3.8]
Statistical Analysis 6: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for social functioning; Test type: Superiority or Other; p = 0.9615, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-3.4 to 3.5]

12. Secondary Outcome: Change From Baseline Between Treatment Comparison in EORTC QLQ-C30 Symptom Scale Scores
Description: as for outcome 11
Time Frame: From Cycle 1 to 14, as of 05 December 2014.
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 335 | 166
Units on a scale
  Fatigue | 1.8 (26.12) [0.1 to 3.5] | 3.3 (24.82) [0.9 to 5.8]
  Nausea and vomiting | 1.7 (26.06) [0.4 to 3.0] | 4.2 (19.71) [2.3 to 6.1]
  Pain | -3.3 (29.02) [-5.1 to -1.5] | 2.0 (30.04) [-0.6 to 4.6]
  Dyspnoea | 2.8 (30.32) [1.0 to 4.7] | 3.3 (24.98) [0.6 to 6.0]
  Insomnia | -2.4 (29.81) [-4.4 to -0.4] | -0.4 (29.30) [-3.3 to 2.5]
  Appetite loss | 1.1 (36.43) [-0.8 to 3.1] | 1.7 (29.61) [-1.1 to 4.6]
  Constipation | 3.5 (32.05) [1.7 to 5.3] | 2.8 (26.05) [0.1 to 5.4]
  Diarrhoea | 1.9 (18.97) [0.6 to 3.1] | 2.4 (26.12) [0.5 to 4.3]
  Financial difficulties | -3.7 (28.87) [-5.6 to -1.9] | -4.0 (26.30) [-6.7 to -1.3]
Statistical Analysis 1: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for fatigue; Test type: Superiority or Other; p = 0.3200, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-4.5 to 1.5]
Statistical Analysis 2: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for nausea and vomiting; Test type: Superiority or Other; p = 0.0369, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-4.8 to -0.2]
Statistical Analysis 3: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for pain; Test type: Superiority or Other; p = 0.0011, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -5.3, 95% CI 2-sided [-8.5 to -2.1]
Statistical Analysis 4: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for dyspnoea; Test type: Superiority or Other; p = 0.7699, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-3.7 to 2.8]
Statistical Analysis 5: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for insomnia; Test type: Superiority or Other; p = 0.2721, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-5.5 to 1.6]
Statistical Analysis 6: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for appetite loss; Test type: Superiority or Other; p = 0.7334, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-4.1 to 2.9]
Statistical Analysis 7: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for constipation; Test type: Superiority or Other; p = 0.6491, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-2.5 to 3.9]
Statistical Analysis 8: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for diarrhoea; Test type: Superiority or Other; p = 0.6293, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.8 to 1.7]
Statistical Analysis 9: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for financial difficulties; Test type: Superiority or Other; p = 0.8812, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-3.1 to 3.6]

13. Secondary Outcome: Change From Baseline Between Treatment Comparison in European Organization for Research and Treatment of Cancer Breast Cancer Module (EORTC QLQ BR23) Functional Scale Scores
Description: The EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of four functional scales (body image, sexual functioning, sexual enjoyment, future perspective) and four symptom scales (systemic side effects, breast symptoms, arm symptoms, upset by hair loss). QLQ-BR23 questionnaire employs 4-point scales with responses from 'not at all' to 'very much'. All scores are converted to a 0 to 100 scale. For functional scales, higher scores represent a better level of functioning.
Time Frame: From Cycle 1 to 14, as of 05 December 2014.
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 335 | 166
Units on a scale
  Body image | 1.9 (28.07) [0.2 to 3.6] | -0.3 (20.33) [-2.8 to 2.1]
  Sexual functioning | -1.1 (16.08) [-2.5 to 0.2] | -0.4 (18.23) [-2.3 to 1.5]
  Sexual enjoyment | -5.2 (20.80) [-8.3 to -2.1] | -6.6 (25.49) [-11.6 to -1.7]
  Future perspective | 8.1 (30.63) [5.8 to 10.4] | 4.5 (30.00) [1.2 to 7.9]
Statistical Analysis 1: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for body image; Test type: Superiority or Other; p = 0.1386, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-0.7 to 5.2]
Statistical Analysis 2: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for sexual functioning; Test type: Superiority or Other; p = 0.5235, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-3.1 to 1.6]
Statistical Analysis 3: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for sexual enjoyment; Test type: Superiority or Other; p = 0.6271, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-4.4 to 7.3]
Statistical Analysis 4: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for future perspective; Test type: Superiority or Other; p = 0.0845, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [-0.5 to 7.6]

14. Secondary Outcome: Change From Baseline Between Treatment Comparison in EORTC QLQ BR23 Symptom Scale Scores
Description: The EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of four functional scales (body image, sexual functioning, sexual enjoyment, future perspective) and four symptom scales (systemic side effects, breast symptoms, arm symptoms, upset by hair loss). QLQ-BR23 questionnaire employs 4-point scales with responses from 'not at all' to 'very much'. All scores are converted to a 0 to 100 scale. For symptom-oriented scales, a higher score represent more severe symptoms.
Time Frame: From Cycle 1 to 14, as of 05 December 2014.
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 335 | 166
Units on a scale
  Systemic therapy side effects | 3.8 (15.19) [2.6 to 4.9] | 3.4 (14.31) [1.8 to 5.0]
  Breast symptoms | -2.2 (21.32) [-3.2 to -1.3] | -1.3 (17.49) [-2.7 to 0.0]
  Arm symptoms | -2.2 (20.59) [-3.6 to -0.9] | -2.0 (20.08) [-4.0 to -0.1]
  Upset by hair loss | 2.9 (30.19) [-1.7 to 7.4] | -6.0 (20.91) [-12.3 to 0.3]
Statistical Analysis 1: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for systemic therapy side effects; Test type: Superiority or Other; p = 0.7273, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.6 to 2.3]
Statistical Analysis 2: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for breast symptoms; Test type: Superiority or Other; p = 0.2671, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-2.6 to 0.7]
Statistical Analysis 3: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for arm symptoms; Test type: Superiority or Other; p = 0.8750, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.6 to 2.2]
Statistical Analysis 4: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Statistical significance for palbociclib plus fulvestrant vs placebo plus fulvestrant for upset by hair loss; Test type: Superiority or Other; p = 0.0255, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 8.9, 95% CI 2-sided [1.1 to 16.6]

15. Secondary Outcome: Change From Baseline Between Treatment Comparison in EuroQoL 5D (EQ-5D)- Health Index Scores
Description: The EuroQol-5D (version 3L) is a brief self-administered, validated instrument consisting of 2 parts. The first part consists of 5 descriptors of current health state (mobility, self care, usual activities, pain/discomfort, and anxiety/ depression); a participant is asked to rate each state on a three level scale (1=no problem, 2=some problem, and 3=extreme problem) with higher levels indicating greater severity/ impairment Published weights are available that allow for the creation of a single summary score called the EQ-5D index, which basically ranges from 0 to 1 with low scores representing a higher level of dysfunction and 1 as perfect health. The second part consists of the EQ-5D general health status as measured by a visual analog scale (EQ-5D VAS). EQ-5D VAS measures the participant's self-rated health status on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: From Cycle 1 to 14, as of 05 December 2014.
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 335 | 166
Units on a scale | 0.006 [-0.01 to 0.03] | -0.031 [-0.06 to 0.00]
Statistical Analysis 1: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Analysis based on repeated measures mixed-effects model with an intercept term, treatment, time, treatment-by-time, and baseline as covariate; Test type: Superiority or Other; p = 0.0308, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.037, 95% CI 2-sided [0.00 to 0.07]

16. Secondary Outcome: Change From Baseline Between Treatment Comparison in EQ-5D Visual Analog Scale (VAS) Scores Scale
Description: The EuroQol-5D (version 3L) is a brief self-administered, validated instrument consisting of 2 parts. The second part consists of the EQ-5D general health status as measured by a visual analog scale (EQ-5D VAS). EQ-5D VAS measures the participant's self-rated health status on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: From Cycle 1 to 14, as of 05 December 2014.
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 335 | 166
Units on a scale | -1.8 (19.00) [-3.3 to -0.3] | -2.6 (23.09) [-4.8 to -0.4]
Statistical Analysis 1: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.5523, Mixed Model Analysis (2-sided) — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-1.9 to 3.5]

17. Secondary Outcome: Time to Deterioration (TTD)
Description: A time to event analysis was pre-specified for pain. An analysis of TTD in pain defined as time between baseline and first occurrence of increase of ≥10 points in pain. Deterioration will be defined increase in score of 10 points or greater from baseline. The Kaplan-Meier estimates of quartiles (time to deterioration) with 95% CI is mentioned below.
Time Frame: Baseline, Day 1 of Cycles 2 to 4, Day 1 of every alternate cycle after that until the end of treatment, as of 05 December 2014
Population: The PRO -evaluable population is defined as a subset of ITT participants, who have completed a baseline and at least one post -baseline PRO assessment prior to end of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 335 | 166
Months
  25% quartile | 1.9 [1.2 to 2.2] | 1.0 [1.0 to 1.9]
  50% quartile | 8.0 [5.6 to NA] — Due to less follow-up time and insufficient number of participants with events. | 2.8 [2.3 to 5.4]
Statistical Analysis 1: Comparison: Palbociclib + Fulvestrant vs Placebo + Fulvestrant; Treatment with palbociclib plus fulvestrant significantly delayed TTD in pain symptom compared with placebo plus fulvestrant for unstratified analysis; Test type: Superiority or Other; p < 0.001, Unstratified log-rank test (1-sided) — The priori threshold for statistical significance is 1-sided alpha=0.025. The p-value was not adjusted for multiple comparisons; 1-sided p-value from the unstratified log-rank test; Hazard Ratio (HR) = 0.642, 95% CI 2-sided [0.487 to 0.846] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs; All Causalities)
Description: An AE is any untoward medical occurrence in a clinical investigation patient administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. An SAE is any untoward medical occurrence at any dose that results in death; is life-threatening; requires hospitalization; results in persistent or significant disability or in congenital anomaly/birth defect. Severity will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.0.
Time Frame: From the date of randomization up to 28 calendar days (±7 days) after last dose of study intervention (up to 8.4 years).
Population: The as-treated (AT) population or safety analysis set included all participants who received at least 1 dose of study intervention, with treatment assignments designated according to actual study intervention received.
Measure: Number; unit: percentage of participants
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 345 | 172
percentage of participants
  With AEs | 98.8 | 93.6
  With SAEs | 22.6 | 19.2
  With Grade 3 or 4 AEs | 80.6 | 26.7
  With Grade 5 AEs | 2.3 | 1.7
  Discontinued palbociclib/placebo due to AEs | 7.5 | 4.7

19. Secondary Outcome: Participants With Shifts From CTCAE Grade ≤2 at Baseline to CTCAE Grade 3 or 4 Postbaseline for Hematology Results
Description: Number of participants with shifts from Grade ≤2 at baseline values to post-baseline values (shift to Grade 3 or 4) were reported as per NCI-CTCAE, V4.0 graded from Grade 1 to 5. Grade 1: Mild; asymptomatic/ mild symptoms; clinical/diagnostic observations only; intervention not indicated. Grade 2: Moderate; minimal, local/noninvasive intervention indicated. Grade 3: Severe/medically significant but not immediately life-threatening; hospitalization/prolongation of hospitalization indicated. Grade 4: Life-threatening consequences; urgent intervention indicated. Shifts in lab parameter from Grade ≤2 at baseline to Grade 3 or 4 postbaseline (for parameters Anemia, Hemoglobin increased, Neutrophil count decreased, Platelet count decreased, and White blood cell count decreased) were reported.
Time Frame: From baseline to end of treatment/withdrawal (up to 4.5 years)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 345 | 172
Participants
  Anemia: number analyzed (Participants) | 343 | 171
  Anemia | 16 | 3
  Hemoglobin increased: number analyzed (Participants) | 343 | 171
  Hemoglobin increased | 1 | 0
  Neutrophil count decreased: number analyzed (Participants) | 342 | 171
  Neutrophil count decreased | 239 | 1
  Platelet count decreased: number analyzed (Participants) | 343 | 171
  Platelet count decreased | 10 | 0
  White blood cell count decreased: number analyzed (Participants) | 343 | 171
  White blood cell count decreased | 167 | 0

20. Secondary Outcome: Participants With Shifts From CTCAE Grade ≤2 at Baseline to CTCAE Grade 3 or 4 Postbaseline for Chemistry Results
Description: Number of participants with shifts from Grade ≤2 at baseline values to post-baseline values (shift to Grade 3 or 4) were reported as per NCI-CTCAE, V4.0 graded from Grade 1 to 5. Grade 1: Mild; asymptomatic/ mild symptoms; clinical/diagnostic observations only; intervention not indicated. Grade 2: Moderate; minimal, local/noninvasive intervention indicated. Grade 3: Severe/medically significant but not immediately life-threatening; hospitalization/prolongation of hospitalization indicated. Grade 4: Life-threatening consequences; urgent intervention indicated. Shifts in lab parameter from Grade ≤2 at baseline to Grade 3 or 4 postbaseline (for parameters ALT increased, ALP increased, AST increased, Blood bilirubin increased, Creatinine increased, Hypercalcemia, Hyperkalemia, Hypermagnesemia, Hypernatremia, Hypoalbuminemia, Hypocalcemia, Hypokalemia, Hypomagnesemia, and Hyponatremia) were reported.
Time Frame: From baseline to end of treatment/withdrawal (up to 4.5 years)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 345 | 172
Participants
  ALT increased: number analyzed (Participants) | 343 | 172
  ALT increased | 10 | 1
  ALP increased: number analyzed (Participants) | 343 | 172
  ALP increased | 2 | 2
  AST increased: number analyzed (Participants) | 343 | 170
  AST increased | 13 | 7
  Blood bilirubin increased: number analyzed (Participants) | 343 | 172
  Blood bilirubin increased | 2 | 3
  Creatinine increased: number analyzed (Participants) | 343 | 172
  Creatinine increased | 5 | 0
  Hypercalcemia: number analyzed (Participants) | 343 | 172
  Hypercalcemia | 1 | 0
  Hyperkalemia: number analyzed (Participants) | 343 | 172
  Hyperkalemia | 2 | 2
  Hypermagnesemia: number analyzed (Participants) | 342 | 172
  Hypermagnesemia | 7 | 2
  Hypernatremia: number analyzed (Participants) | 343 | 172
  Hypernatremia | 0 | 1
  Hypoalbuminemia: number analyzed (Participants) | 342 | 171
  Hypoalbuminemia | 0 | 1
  Hypocalcemia: number analyzed (Participants) | 343 | 172
  Hypocalcemia | 2 | 2
  Hypokalemia: number analyzed (Participants) | 343 | 172
  Hypokalemia | 0 | 0
  Hypomagnesemia: number analyzed (Participants) | 342 | 171
  Hypomagnesemia | 0 | 0
  Hyponatremia: number analyzed (Participants) | 343 | 172
  Hyponatremia | 12 | 4

ADVERSE EVENTS:
Time Frame: From the date of randomization up to 28 calendar days (±7 days) after last dose of study intervention (up to 8.4 years).
Description: The safety analysis set for adverse events and serious adverse events included all participants who received at least 1 dose of study intervention, with treatment assignments designated according to actual study intervention received.
  All-cause mortality of the total number at risk included all participants who were randomized, with study intervention, regardless of whether participants received the study intervention or received a different drug from that to which they were randomized.
Arm/Group | Palbociclib + Fulvestrant | Placebo + Fulvestrant
All-Cause Mortality (participants affected / at risk) | 201/347 | 109/174
Serious Adverse Events (participants affected / at risk) | 78/345 | 33/172
Other Adverse Events (participants affected / at risk) | 341/345 | 161/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Fulvestrant (N=345) | Placebo + Fulvestrant (N=172)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 2
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Disease progression (General disorders) | 4 | 0
General physical health deterioration (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 5 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 3 | 2
Pyelonephritis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Drug withdrawal convulsions (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric volvulus (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hiatus hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Injection site fibrosis (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Heat illness (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Sedation complication (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0
Device occlusion (Product Issues) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Facial spasm (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Vocal cord paresis (Nervous system disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Fulvestrant (N=345) | Placebo + Fulvestrant (N=172)
Anaemia (Blood and lymphatic system disorders) | 108 | 23
Leukopenia (Blood and lymphatic system disorders) | 113 | 2
Neutropenia (Blood and lymphatic system disorders) | 231 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 51 | 0
Abdominal pain (Gastrointestinal disorders) | 31 | 13
Constipation (Gastrointestinal disorders) | 77 | 29
Diarrhoea (Gastrointestinal disorders) | 95 | 35
Dry mouth (Gastrointestinal disorders) | 27 | 16
Dyspepsia (Gastrointestinal disorders) | 41 | 9
Nausea (Gastrointestinal disorders) | 126 | 51
Stomatitis (Gastrointestinal disorders) | 51 | 5
Vomiting (Gastrointestinal disorders) | 76 | 27
Asthenia (General disorders) | 27 | 14
Chest pain (General disorders) | 16 | 11
Fatigue (General disorders) | 151 | 56
Injection site pain (General disorders) | 26 | 19
Oedema peripheral (General disorders) | 36 | 13
Pain (General disorders) | 20 | 14
Pyrexia (General disorders) | 44 | 9
Nasopharyngitis (Infections and infestations) | 50 | 14
Upper respiratory tract infection (Infections and infestations) | 46 | 13
Aspartate aminotransferase increased (Investigations) | 42 | 13
Neutrophil count decreased (Investigations) | 84 | 2
Platelet count decreased (Investigations) | 43 | 0
White blood cell count decreased (Investigations) | 107 | 7
Decreased appetite (Metabolism and nutrition disorders) | 61 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 90 | 42
Back pain (Musculoskeletal and connective tissue disorders) | 65 | 32
Muscle spasms (Musculoskeletal and connective tissue disorders) | 35 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 21 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 35 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 62 | 27
Dizziness (Nervous system disorders) | 59 | 18
Dysgeusia (Nervous system disorders) | 18 | 5
Headache (Nervous system disorders) | 102 | 38
Anxiety (Psychiatric disorders) | 20 | 10
Depression (Psychiatric disorders) | 27 | 10
Insomnia (Psychiatric disorders) | 46 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 79 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 50 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 25 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 53 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 68 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 32 | 14
Rash (Skin and subcutaneous tissue disorders) | 46 | 8
Hot flush (Vascular disorders) | 57 | 30
Lacrimation increased (Eye disorders) | 27 | 2
Vision blurred (Eye disorders) | 23 | 3
Abdominal distension (Gastrointestinal disorders) | 21 | 9
Abdominal pain upper (Gastrointestinal disorders) | 24 | 15
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 23 | 3
Influenza like illness (General disorders) | 34 | 5
Influenza (Infections and infestations) | 12 | 10
Urinary tract infection (Infections and infestations) | 38 | 14
Contusion (Injury, poisoning and procedural complications) | 20 | 4
Fall (Injury, poisoning and procedural complications) | 18 | 13
Alanine aminotransferase increased (Investigations) | 32 | 9
Blood alkaline phosphatase increased (Investigations) | 13 | 11
Blood creatinine increased (Investigations) | 20 | 3
Weight decreased (Investigations) | 18 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 28 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 18 | 8
Paraesthesia (Nervous system disorders) | 19 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 29 | 3
Hypertension (Vascular disorders) | 26 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-10-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT01942135/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT01942135/SAP_001.pdf